CLINICAL TRIAL: NCT06441461
Title: Mental Health and Occupational Outcomes Among Informal Caregivers at Work - a Danish Nationwide Register-based Cohort Study
Brief Title: Informal Caregivers at Work - Phase 2
Acronym: PPJob-II
Status: Active, not recruiting | Type: Observational
Sponsor: Team Working Life Denmark (Industry)
Collaborators: Bispebjerg Hospital (Other); Herlev and Gentofte Hospital (Other); HMW Health and Communication (Unknown); National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Sponsor
Other Study IDs: TeamWorkingLifeDenmark
Record Dates: First submitted 2024-05-21; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Work-Related Stress
Keywords: Mental health issue; Work-related illness; Loss of career progression
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish citizens: All citizens aged 0-25 years and all adults aged 18-67 years residing in Denmark in the period from 2000 to 2008.
  Interventions: Other: Primary informal caregiver at work.

INTERVENTIONS:
Other: Primary informal caregiver at work. — Employees becoming a primary informal caregiver for a child or an adolescent with mental health problems in the period from 2000 to 2018.

SUMMARY:
Mental health problems are rising among children and adolescents. This may not only impact the child's level of daily functioning but also close family members. Informal caregiving is defined as unpaid care for a sick, disabled, or other closely related person. Providing long-term informal care has been associated with detrimental stress-related outcomes, and being simultaneously active in the labor market has been highlighted as an increased burden for the caregiver. Workplaces are poorly suited for dealing with private stressors despite their potential negative consequences for the caregiver's job status and health. There is a need for improving understanding of how long-term informal caregiving impacts job and health outcomes, as well as for measures minimizing potential negative consequences among at-risk occupational groups.

DETAILED DESCRIPTION:
This Danish nationwide observational cohort study examines the associations between employees being a primary informal caregiver for a child or adolescent with mental health problems and the employees' occupational and health outcomes. In addition, we seek to identify modifying psychosocial risk factors at work as well as at-risk occupational groups. The study relies on pre-existing longitudinal data extracted from Danish national registers, including highly reliable information on occupational status, birth information, residence, public transfer payments, income, psychiatric treatment and services, treatment for substance abuse, psychotropic prescription drugs redeemed, as well as background information. In Denmark, all citizens are assigned with a unique identification number enabling merging of national register data included. Caregiver-child relationships are established based on merging of data from birth and household registers. In this study, register data are further merged with information on psychosocial work environment based on national survey data. All data are located at Statistics Denmark, and accessed and analyzed via a logged, secured platform, The Danish Occupational Cohort (DOC*X) (www.DOC-X.dk). Exposed employees are compared to a reference group of employees without mental health problems at the familiy level matched according to age group, gender (female/male), and socio-occupational status.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents: Citizens aged 0-25 years in the period between 2000 and 2018. Mental disorder is indicated by redeeming of psychotropic medication, treatment for substance abuse, and psychiatric services. Children of reference adult caregivers is defined by having no personal history of a mental disorder. We exclude children born outside of Denmark.
* Adults: Citizens aged 18-67 years residing in Denmark, partaking in the work force in the period between 2000-2008, and living with a child in the household at any time until the child's 18th year or being a parent to a child at its birth.

Exclusion Criteria:

* We exclude all citizens born in the Faroe Islands and in Greenland. We exclude all citizens residing in the Faroe Islands and in Greenland in the period between 2000 and 2018.

Ages: 0 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a nationalwide register-based study of occupational and mental health outcomes of all adult caregivers to children with and without mental health problems.
Sampling Method: Non-Probability Sample
Enrollment: 4386647 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Personal gross income (Level of analysis: primary informal caregiver) | Up to 10 years of follow-up.
  Personal gross income is analyzed as series of annual statuses.
Employment (Level of analysis: primary informal caregiver). | Up to 10 years of follow-up.
  Employment is analyzed as series of annual statuses (i.e., number of weeks employed within each year during follow-up).
Long-term sickness absence (Level of analysis: primary informal caregiver). | Up to 10 years of follow-up.
  Long-term sickness absence is analyzed as time-to-event from baseline on the week scale.
Mental health (Level of analysis: primary informal caregiver). | Up to 10 years of follow-up.
  Mental health is analyzed as time-to-event from baseline on the week scale whichever comes first: redeemed psychotropic drug prescriptions, treatment for substance abuse or psychiatric hospital services.

SECONDARY OUTCOMES:
Moderation of potential associations by psychosocial work environment (Level of analysis: primary informal caregiver) | JEMs were composed of national survey data collected in 2000 and 2005.
  Moderation of potential association by psychosocial work environment is based on age- and sex-specific job-exposure matrices (JEM).
Moderation of potential associations by occupational group (Level of analysis: primary informal caregiver). | Annual data in the period between 2000 and 2018.
  Moderation by occupational group is based on DISCO-88 codes (International Standard Classification of Occupation, Danish version 1988).

CONTACTS AND LOCATIONS:
Overall Officials: Johan H Jensen, PhD, Principal Investigator — Team Working Life Denmark; Johan H Jensen, PhD, Principal Investigator — Occupational and Environmental Medicine, Copenhagen University Hospital - Bispebjerg & Frederiksberg
Locations (1):
- Team Working Life Denmark, Valby, Denmark

IPD SHARING:
Plan to Share IPD: No
Statistics Denmark's extensive collections of registers contain a significant potential for research and analysis.
  In order to use this research and analysis potential in accordance with the current register legislation and Statistics Denmark's data confidentiality principles, Statistics Denmark has established special micro-data schemes (Research Scheme, Authority Scheme and Legislative Model).
  Through the micro-data schemes, microdata (i.e. individual/single company data) is made available for specific research, investigation and analysis tasks for authorised research/analysis environments. Foreign research/analysis environments cannot be authorised for the scheme, but under certain conditions, foreign users can access data.
  Further information: https://www.dst.dk/en/TilSalg/Forskningsservice/Dataadgang